CLINICAL TRIAL: NCT03204734
Title: Evaluate Effectiveness and Security of Capecitabine or Endocrinotherapy as a Maintenance Therapy Regimen After 2nd-line or Over 2nd-line Therapy With Capecitabine Combine Regimen in Hormone Receptor Positive and HER2 Negative Metastatic Breast Cancer
Brief Title: Capecitabine or Endocrinotherapy as a Maintenance Therapy Regimen at Least 2nd Line in Hormone Receptor Positive and HER2 Negative Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhengyabing, Chief Physician, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH15009
Record Dates: First submitted 2017-06-24; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: therapy; Capecitabine; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capecitabine (Experimental): Capecitabine by mouth twice per day for 14 days, per 21 days as a cycle, until disease progress or toxicity can not be tolerated.Capecitabine starting dose was the dose used at the end of the combined chemotherapy regimen,eg:1000mg per BSA.
  Interventions: Drug: Capecitabine
- endocrine therapy (Experimental): endocrine therapy will been given as a sequential treatment in Metastatic breast cancer patients who are got benefit in capecitabine-base chemotherapy.The medicine will be confirmed by the patient's past-treatment.
  Interventions: Drug: endocrine therapy

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will been given as a sequential treatment who are got benefit in capecitabine-base chemotherapy.
  Arms: Capecitabine
Drug: endocrine therapy — endocrine therapy will been given as a sequential treatment who are got benefit in capecitabine-base chemotherapy.Endocrine therapy is determined by the doctor, including any kind of letrozole, anastrozole, exemestane, fulvestrant, tamoxifen, toremifene, combined with or without drugs or surgery in the inhibition of ovarian function.
  Arms: endocrine therapy

SUMMARY:
A single-site study about the efficacy of sequential monotherapy: Capecitabine vs. endocrine therapy, in metastatic breast cancer patients with HR-positive & HER2-negative after capecitabine-base chemotherapy.

DETAILED DESCRIPTION:
Capecitabine-base chemotherapy must be ≥Second-line Therapy

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* The age is Above 18 years of age, <70 years old
* HR-positive & HER2-negative
* Metastatic breast cancer,incurable.
* For recurrent or metastatic lesions has had at least 1 but no more than 3 kinds of chemotherapy, if there is disease progression within 6 months after the end of the adjuvant chemotherapy, adjuvant chemotherapy will been the first-line treatment for metastatic lesions
* No prior use of capecitabine therapy or the use of capecitabine treatment was effective, and the efficacy evaluation was CR/PR/SD more than 6 months.
* Eastern Cooperative Oncology Group performance status (ECOG PS)=0~1
* The basic function of normal bone marrow
* Functions of liver and kidney is normal
* Expectation of life is more than 3 months
* Agreed to take contraceptive measures during treatment

Exclusion Criteria:

* Previous toxicity was not recovered to 0-1 degrees
* Central nervous system metastasis
* Pregnancy or lactation
* There are uncontrolled infection, myocardial infarction, thrombosis, etc.
* There are uncontrolled chronic diseases such as diabetes, hypertension, peptic ulcer, chronic hepatitis, mental disease;
* Researchers believe that is not suitable for the study
* Patients with other malignant tumor history, except the healed skin basal cell carcinoma and carcinoma of uterine cervix;
* Bilateral breast cancer
* Capecitabine was ineffective in past treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | From date of enrolling until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  Progression-free survival (PFS) is defined as the time elapsed between enrolling and tumor progression or death from any cause

SECONDARY OUTCOMES:
clinical benefit rate(CBR) | From date of enrolling until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  the response is CR+PR+SD ≥ 24 weeks
overall survival | From date of enrolling until the date of death from any cause, assessed up to 3 years
  the time elapsed between enrolling and death from any cause
Number of participants with Grade 3/4 adverse events | From date of enrolling until the date of 1 month of stop treatment, assessed up to 3 years
  Number of Participants with Grade 3/4 Adverse Events
Quality of life(QOL)（1） | From date of enrolling until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  change from enrolling to progression disease or death according EORTC QLQ-C30
Quality of life(QOL)（2） | From date of enrolling until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  change from enrolling to progression disease or death according EORTC BR23

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-jia Wang, PHD,MD, Principal Investigator — Zhejiang Cance Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muss HB, Case LD, Richards F 2nd, White DR, Cooper MR, Cruz JM, Powell BL, Spurr CL, Capizzi RL. Interrupted versus continuous chemotherapy in patients with metastatic breast cancer. The Piedmont Oncology Association. N Engl J Med. 1991 Nov 7;325(19):1342-8. doi: 10.1056/NEJM199111073251904. PMID 1922236